CLINICAL TRIAL: NCT05858099
Title: The Early Detection and Progression of Subclinical Atherosclerosis in Psoriasis (EDSAP): Protocol for an Observational, Prospective Cohort Study
Brief Title: The Early Detection and Progression of Subclinical Atherosclerosis in Psoriasis
Acronym: EDSAP
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: HM Sanchinarro University Hospital (Other); Hospital Universitario 12 de Octubre (Other); Medstar Health Research Institute (Other); Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Principal Investigator, Alvaro Gonzalez Cantero, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: CI-BIOB-058-01
Record Dates: First submitted 2023-04-12; First posted 2023-05-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis; Atherosclerosis
Keywords: Imaging; Inflammation; Coronary computed tomography angiography; Biomarkers; Cardiovascular disease; Molecular biomarkers
MeSH Terms: conditions — Psoriasis; Atherosclerosis; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify new molecular and imaging markers associated with the presence of atherosclerosis and its progression in psoriasis. The main questions it aims to answer are:

* To assess the prevalence, vascular distribution and burden of subclinical atherosclerosis in patients with psoriasis and its relationship with inflammatory biomarkers and cardiovascular (CV) risk algorithms using 2D vascular ultrasound (2DVUS) of carotid and femoral arteries, 3D vascular ultrasound (3DVUS) of carotid and femoral arteries and Coronary Computed Tomography Angiography (CCTA).
* To characterize the composition of atherosclerotic plaques by CCTA and 3DVUS of the carotid and femoral arteries.
* To evaluate the effect of different treatments used in psoriasis on the progression and characterisation of subclinical atherosclerosis in different arterial territories assessed by non-invasive imaging techniques.
* To characterise the atherosclerosis process in patients with psoriasis using laboratory analysis and "-omics" technologies, as well as to evaluate changes at the molecular level after treatment of the skin disease.

Participants will undergo 2 study visits:

* At baseline, before starting biologic treatment for psoriasis. A 1-year follow up, after having completed one year under biologic treatment for psoriasis.
* Both visits include a clinical interview, physical examination, fasting blood draw and assessment of atherosclerotic disease by non-invasive vascular imaging tests (2D/3DVUS and CCTA).
* Participants may undergo an unscheduled clinical visit if the patient suffers a worsening of the psoriasis. This visit includes a clinical interview, physical examination and fasting blood draw.

DETAILED DESCRIPTION:
Life expectancy of patients with psoriasis is reduced by 4-5 years due to cardiovascular (CV) disease with an increased risk of myocardial infarction at an earlier age compared to general population. This increased risk is independent of traditional CV risk factors and higher in moderate-to-severe forms of psoriasis. Inflammation may play a key role in the development of atherosclerosis in these patients. The EDSAP study aims to identify new molecular and imaging markers associated with the presence of atherosclerosis and its progression in a chronic inflammatory state such as psoriasis in order to help improve primary CV prevention strategies, understand the effect of biologic drugs on the CV system and serve as a model for understanding atherosclerosis in other chronic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients eligible for biologic therapy.
* Psoriasis patients aged between 30 to 65 years.

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, angina pectoris, peripheral vascular disease, aortic aneurysm, angioplasty, cardiac surgery, atrial fibrillation or any other cardiological condition).
* Patients undergoing oncological treatment.
* History of transplantation with active immunosuppressive or immunomodulatory treatment.
* Patients with morbid obesity (body mass index ≥40 kg/m2).
* Patients with diabetes mellitus.
* Patients with chronic liver disease.
* Patients with chronic kidney disease (glomerular filtration rate <60 mL/min/1.73 m2).
* Patients with other chronic inflammatory disease, presence of any pathology that decreases life expectancy to less than 3 years, or any disease or condition that could affect adherence to study procedures.
* Patients that have had a chest computed tomography scan in the previous year.
* Pregnant or breastfeeding women.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients diagnosed with psoriasis clinically by an expert physician and deemed suitable for biologic therapy by the investigator
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of subclinical coronary artery atherosclerosis in patients with psoriasis by CCTA | 4-6 years
  To determine presence / absence of atheroma plaques in the coronary artery by CCTA
Prevalence of subclinical atherosclerosis in carotid and femoral arteries of patients with psoriasis by 2DVUS | 4-6 years
  To determine presence / absence of atheroma plaques by 2DVUS for femoral and carotid arteries.

SECONDARY OUTCOMES:
CCTA Quantitative Assessment of plaques by plaque volume (mm3) | 4-6 years
  To quantitatively assess atheroma plaques from the coronary artery by CCTA, measured in mm3
Carotid and femoral 3DVUS quantitative plaque assessment by plaque volume (mm3) | 4-6 years
  Quantitatively assess atheroma plaques in the femoral and carotid arteries by 3DVUS, measured in mm3.
Proteomic signature characterization by Liquid Chromatography- Mass Spectrometry (LC-MS/MS) | 4-6 years
  To characterize potential proteomic biomarkers by LC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Álvaro González Cantero, MD, PhD, Principal Investigator — Fundación Hospital Ramón y Cajal
Locations (1):
- Ramón y Cajal University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abbad-Jaime de Aragon C, Berna-Rico E, Ballester-Martinez MA, Jaen P, Solis J, Barderas MG, Fernandez-Friera L, N Mehta N, Gelfand JM, Gonzalez-Cantero A. Early Detection and Progression of Subclinical Atherosclerosis in Psoriasis (EDSAP): protocol for an observational, single-centre, prospective cohort study. BMJ Open. 2023 Sep 26;13(9):e072455. doi: 10.1136/bmjopen-2023-072455. PMID 37751953